CLINICAL TRIAL: NCT06598397
Title: Using Multiphase Optimization Strategy (MOST) to Optimize a Cost-effective, Sustainable and Scalable Smoking Cessation Package for Smokers in HIV Clinical Care
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CA268932
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-10

CONDITIONS: Human Immunodeficiency Virus (HIV); Smoking Cessation
Keywords: MOST; multiphase optimization strategy; implementation; HIV clinical care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Smoking Cessation | interventions — Motivational Interviewing; Counseling

STUDY DESIGN:
Intervention Model Description: A full factorial randomized controlled trial using Multiphase Optimization STrategy (MOST) with 4 component interventions, each at 2 levels (off/on), for a total of 16 component conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (16):
- Condition 1 (No Intervention): Participants will receive the Core Component.
- Condition 2 (Experimental): Participants will receive the Core Component and Combination-NRT intervention.
  Interventions: Drug: Combination NRT
- Condition 3 (Experimental): Participants will receive the Core Component and Text Messaging intervention.
  Interventions: Behavioral: Skills-based Text Messaging
- Condition 4 (Experimental): Participants will receive the Core Component as well as the Combination-NRT and Text Messaging interventions.
  Interventions: Behavioral: Skills-based Text Messaging; Drug: Combination NRT
- Condition 5 (Experimental): Participants will receive the Core Component and Peer Mentoring intervention.
  Interventions: Behavioral: Peer Mentoring
- Condition 6 (Experimental): Participants will receive the Core Component as well as the Combination-NRT and Peer Mentoring interventions.
  Interventions: Behavioral: Peer Mentoring; Drug: Combination NRT
- Condition 7 (Experimental): Participants will receive the Core Component as well as the Text Messaging and Peer Mentoring interventions.
  Interventions: Behavioral: Peer Mentoring; Behavioral: Skills-based Text Messaging
- Condition 8 (Experimental): Participants will receive the Core Component as well as the Combination-NRT, Text Messaging and Peer Mentoring interventions.
  Interventions: Behavioral: Peer Mentoring; Behavioral: Skills-based Text Messaging; Drug: Combination NRT
- Condition 9 (Experimental): Participants will receive the Core Component and Motivational Interviewing Counseling intervention.
  Interventions: Behavioral: Motivational Interviewing (MI) Counseling
- Condition 10 (Experimental): Participants will receive the Core Component as well as the Combination-NRT and Motivational Interview Counseling interventions.
  Interventions: Behavioral: Motivational Interviewing (MI) Counseling; Drug: Combination NRT
- Condition 11 (Experimental): Participants will receive the Core Component as well as the Text Messaging and Motivational Interview Counseling interventions.
  Interventions: Behavioral: Motivational Interviewing (MI) Counseling; Behavioral: Skills-based Text Messaging
- Condition 12 (Experimental): Participants will receive the Core Component as well as the Combination-NRT, Text Messaging and Motivational Interview Counseling interventions.
  Interventions: Behavioral: Motivational Interviewing (MI) Counseling; Behavioral: Skills-based Text Messaging; Drug: Combination NRT
- Condition 13 (Experimental): Participants will receive the Core Component as well as the Peer Mentoring and Motivational Interview Counseling interventions.
  Interventions: Behavioral: Motivational Interviewing (MI) Counseling; Behavioral: Peer Mentoring
- Condition 14 (Experimental): Participants will receive the Core Component as well as the Combination-NRT, Peer Mentoring and Motivational Interview Counseling interventions.
  Interventions: Behavioral: Motivational Interviewing (MI) Counseling; Behavioral: Peer Mentoring; Drug: Combination NRT
- Condition 15 (Experimental): Participants will receive the Core Component as well as the Text Messaging, Peer Mentoring and Motivational Interview Counseling interventions.
  Interventions: Behavioral: Motivational Interviewing (MI) Counseling; Behavioral: Peer Mentoring; Behavioral: Skills-based Text Messaging
- Condition 16 (Experimental): Participants will receive the Core Component as well as the Combination-NRT, Text Messaging, Peer Mentoring, and Motivational Interview Counseling interventions.
  Interventions: Behavioral: Motivational Interviewing (MI) Counseling; Behavioral: Peer Mentoring; Behavioral: Skills-based Text Messaging; Drug: Combination NRT

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI) Counseling — Six sessions of phone counseling over 10-12 weeks with MI counselor trained in motivational interviewing and tobacco use treatment.
  Arms: Condition 10; Condition 11; Condition 12; Condition 13; Condition 14; Condition 15; Condition 16; Condition 9
Behavioral: Peer Mentoring — Eight sessions of informal counseling with an experienced peer former smoker living with HIV to model healthy behavior and provide practical advice and tips for quitting based on their lived experience.
  Arms: Condition 13; Condition 14; Condition 15; Condition 16; Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Skills-based Text Messaging — NCI's 8-week text messaging smoking cessation program, smokefreeTXT.gov.
  Arms: Condition 11; Condition 12; Condition 15; Condition 16; Condition 3; Condition 4; Condition 7; Condition 8
Drug: Combination NRT — If they smoke 10 or more cigarettes per day (CPD), participants will receive 2 weeks of 21 mg patches, 2 weeks of 14 mg patches and 2 weeks of 7 mg patches; if they smoke less than 10 CPD, participants will receive 4 weeks of 14 mg patches and 2 weeks of 7 mg patches. Participants will receive either 2 or 4 mg of nicotine lozenges for a total of up to 20 lozenges per day.
  Arms: Condition 10; Condition 12; Condition 14; Condition 16; Condition 2; Condition 4; Condition 6; Condition 8

SUMMARY:
This study's long-term goal is to improve clinical outcomes among smokers living with HIV (SLWH) by providing smoking cessation interventions in HIV clinical care that will increase the chances of quitting smoking, limits costs and burden on staff and reach many smokers living with HIV.

DETAILED DESCRIPTION:
This study will utilize Multiphase Optimization Strategy (MOST) to optimize a smoking cessation treatment for HIV clinical care by directly targeting patient barriers to quitting and clinical care barriers to reaching and effectively treating a broad heterogeneous population of smokers living with HIV. The four intervention components will be aimed at barriers to quitting among smokers living with HIV and include Motivational Interviewing; Peer Mentoring; Text-messaging; Combination Nicotine Replacement Therapy. These components have shown promise in research but are under-utilized to help smokers living with HIV quit and have not been tested in an optimization trial. This study will also incorporate data to evaluate the fidelity, acceptability and feasibility of the interventions in the HIV clinical care context in order to identify the most cost-effective, sustainable and scalable tobacco treatment package for the care environment.

ELIGIBILITY:
Inclusion Criteria:

* Status as HIV+
* Age 18 or older
* Currently smokes ≥ 5 CPD, on average, in past month
* Positive for salivary cotinine
* Able to understand the nature of the study and the consenting process
* Is engaged in HIV clinical care
* Living in larger NYC metropolitan area currently and for the next 6-8 months

Exclusion Criteria:

* Suffers from any medical condition or contraindication precluding use of nicotine replacement therapy
* Current use of any tobacco cessation medications (varenicline, NRT patch, nicotine gum, lozenge, spray or inhaler, or bupropion)
* Currently participating in a smoking cessation program
* Pregnant or nursing and plans to be in next 6 months
* Has schizophrenia/schizo-affective disorder
* Does not have a functioning mobile phone that can receive text messages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Biochemically-validated 7-day point prevalence smoking abstinence among SLWH in HIV clinical care | 24-32 weeks
  Self-reported 7-day cigarette PPA (point prevalence abstinence), with biochemical verification of CO (carbon monoxide) ≤6 ppm and negative salivary cotinine assessment

SECONDARY OUTCOMES:
Self-reported 30-day PPA | 24-32 weeks
  Self-reported 30-day cigarette PPA (point prevalence abstinence), with biochemical verification of CO (carbon monoxide) ≤6 ppm and negative cotinine assessment
Self-reported 7-day PPA | 6-10 and 12-16 weeks
  Self-reported 7-day cigarette PPA (point prevalence abstinence)
Self-reported 30-day PPA | 6-10 and 12-16 weeks
  Self-reported 30-day cigarette PPA (point prevalence abstinence), with biochemical verification of CO (carbon monoxide) ≤6 ppm and negative cotinine assessment
Quit attempts | 6-10, 12-16, and 24-32 weeks
  Number of quit attempts (of at least 24 hours) in last 7 days and since last assessment

CONTACTS AND LOCATIONS:
Locations (1):
- New York University School of Global Public Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No